CLINICAL TRIAL: NCT01387217
Title: A Single-blind, Placebo-controlled, Two Part Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Doses of GSK2018682 in Healthy Volunteers
Brief Title: GSK2018682 FTIH in Healthy Volunteers
Acronym: P1A114070
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 114070
Record Dates: First submitted 2011-04-14; First posted 2011-07-04 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Multiple Sclerosis
Keywords: GSK2018682; First Time in Human; Healthy Volunteer
MeSH Terms: conditions — Multiple Sclerosis | interventions — GSK2018682

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): Part A will be used to confirm the prediction of GSK2018682 PK, assess its effects on lymphocytes, and monitor its safety profile in a single cohort (Cohort 1). Cohort 1 will consist of 4 subjects and explore 4 doses of GSK2018682 in 4 study sessions. In each session, three subjects will receive GSK2018682 and one subject will receive placebo. Thus, when the cohort completes, each subject will receive placebo and 3 doses of GSK2018682.
  Interventions: Drug: GSK2018682; Drug: Placebo
- Part B (Experimental): Part B will explore doses to refine the dose-response curve of GSK2018682 on lymphocyte suppression, as allowed by stopping criteria, in 1 or 2 cohorts of up to 15 subjects (Cohort 2 and Cohort 3). In Part B, up to six single ascending doses of GSK2018682 and one dose of placebo will be investigated in up to 8 sessions.
  Interventions: Drug: GSK2018682; Drug: Placebo

INTERVENTIONS:
Drug: GSK2018682 — GSK2018682
Drug: Placebo — Matched Placebo

SUMMARY:
This protocol describes the first administration of GSK2018682 to humans. The study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of single ascending doses of GSK2018682. The study will also provide preliminary evidence of the potential therapeutic dose-range by measuring the inhibitory effect of GSK2018682 on total lymphocyte counts.

DETAILED DESCRIPTION:
This protocol describes the first administration of GSK2018682 to humans. The study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of single ascending doses of GSK2018682. The study will also provide preliminary evidence of the potential therapeutic dose-range by measuring the inhibitory effect of GSK2018682 on total lymphocyte counts.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters significantly outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Subjects with lymphocyte counts outside the normal range should always be excluded from enrollment
* BMI within the range 19 - 28 kg/m2 (inclusive).

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption
* Subjects with a history of, or examination suspicious for, skin cancer(s) including melanoma, basal cell or squamous cell carcinoma.
* Systolic blood pressure less than 95 mmHg or greater than 140 mmHg, or diastolic blood pressure less than or equal to 50 mmHg or greater than or equal to 95 mmHg.
* Symptomatic reduction in blood pressure after orthostatic challenge.
* Subjects with resting heart rate less than 45 beats per minute or greater than 90 beats per minute

Other criteria may apply as defined by the clinical protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2010-05-21 (Actual); Primary Completion 2010-12-20 (Actual); Study Completion 2010-12-20 (Actual)

PRIMARY OUTCOMES:
To investigate the safety and tolerability of single escalating oral doses of GSK2018682 | Participants will be followed and monitored for the duration of their hospital stay. The longest duration of participation in the study will be approximately 12 weeks
  Adverse event and safety lab monitoring
To investigate effects of GSK2018682 on heart rate and blood pressure | Participants will be followed and monitored for the duration of their hospital stay. The longest duration of participation in the study will be approximately 12 weeks
  12 lead ECG and telemetry monitoring plus vital signs (systolic and diastolic blood blood pressures), heart rate, respiratory rate and temperature
To investigate the pharmacokinetics of single doses of GSK2018682 | Participants will be followed and monitored for the duration of their hospital stay. The longest duration of participation in the study will be approximately 12 weeks
  Peak blood concentration, time of peak blood concentration, oral clearance, half life and AUC
Evaluate the effect of single escalating oral doses of GSK2018682 on lymphocytes (totals plus subsets) | Participants will be followed and monitored for the duration of their hospital stay. The longest duration of participation in the study will be approximately 12 weeks
  Reduction from baseline in lymphocyte counts obtained at different time points after dosing and at different dose levels

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Australia (2):
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 114070 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114070?search=study&search_terms=114070#rs
- Available data/document: Individual Participant Data Set: 114070 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114070 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114070 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114070 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114070 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114070 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114070 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register